CLINICAL TRIAL: NCT02101164
Title: An Open-Label, Multicentre Trial to Evaluate the Time Associated With the Preparation and Administration of Denosumab and Pamidronate in Subjects With Solid Tumors and Metastatic Bone Disease in Canada
Brief Title: Evaluate Time Associated With the Preparation & Administration of Denosumab/Pamidronate in Patients With Solid Tumors and Metastatic Bone Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 20120127
Record Dates: First submitted 2014-03-12; First posted 2014-04-02 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-01

CONDITIONS: Solid Tumor; Metastatic Bone Disease
MeSH Terms: conditions — Bone Diseases | interventions — Denosumab; Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Active Comparator): 1 dose of denosumab every 4 weeks for 2 doses, followed by 1 dose of pamidronate every 4 weeks for 2 doses.
  Interventions: Biological: denosumab; Drug: pamidronate
- Treatment Group B (Active Comparator): 1 dose of pamidronate every 4 weeks for 2 doses, followed by 1 dose of denosumab every 4 weeks for 2 doses.
  Interventions: Biological: denosumab; Drug: pamidronate

INTERVENTIONS:
Biological: denosumab — Treatment Group A - 120 mg SC dose every 4 weeks at Day 1 and week 5 Treatment Group B - 120 mg SC dose every 4 weeks at Week 9 and Week 13
  Other Names: XGEVA
Drug: pamidronate — Treatment Group A - 90 mg IV dose every 4 weeks at Week 9 and Week 13 Treatment Group B - 90 mg IV dose every 4 weeks at Day 1 and Week 5
  Other Names: Aredia

SUMMARY:
This study will estimate the total time for the preparation and administration of denosumab and the total time for the preparation and administration of pamidronate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic bone disease secondary to a solid tumor (eg, breast cancer, lung cancer, etc).
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject is one of the following:

  * being considered for pamidronate IV infusions or denosumab SC injections for treatment of metastatic bone disease (prescribed per Canadian product monograph); OR
  * scheduled to receive pamidronate IV infusions or denosumab SC injections for treatment of metastatic bone disease (prescribed per Canadian product monograph); OR
  * currently receiving pamidronate IV infusions or denosumab SC injections for treatment of metastatic bone disease AND has received no more than 4 prior administration of either product combined (prescribed per Canadian product monograph).
* Subject has a serum calcium or albumin-adjusted serum calcium ≥ 2.0 mmol/L (8.0 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL)

Exclusion Criteria:

* Diagnosis with metastatic bone disease secondary to multiple myeloma or prostate cancer.
* Severe renal impairment (creatinine clearance < 30 mL/min)
* Subject is being considered for ambulatory pamidronate administration using an infuser device (ie, "baby bottle").
* A known active infection with Hepatitis B virus or Hepatitis C virus.
* Subject has known positive results for human immunodeficiency virus (HIV).Subject has a history of other malignancy within the past 5 years, other than:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 5 years before enrollment and felt to be at low risk for recurrence by the treating physician
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated cervical carcinoma in situ without evidence of disease
  * Adequately treated breast ductal carcinoma in situ without evidence of disease
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer
  * Adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ.
* Subject has a history or current evidence of osteonecrosis/osteomyelitis of the jaw, active dental or jaw condition that requires oral surgery, non-healed dental/oral surgery, or planned invasive dental procedure over the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Total duration (in hours, minutes and seconds) for investigational product preparation and administration | Day 1
Total duration (in hours, minutes and seconds) for investigational product preparation and administration | Week 5
Total duration (in hours, minutes and seconds) for investigational product preparation and administration | Week 9
Total duration (in hours, minutes and seconds) for investigational product preparation and administration | Week 13

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com